CLINICAL TRIAL: NCT04354584
Title: Early and Late Pulmonary and Systemic Inflammation in Critically Ill, Mechanically Ventilated Patients With Verified COVID-19
Brief Title: Compartmental Inflammation in Mechanically Ventilated Patients With COVID-19
Acronym: COV2ICU-DK
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ronni R. Plovsing, MD, PhD, Hvidovre University Hospital
Other Study IDs: COV2ICU-DK; H-20023159 (Other: Research Ethical Committee of The Capital Region of Denmark); R349-2020-540 (Other Grant/Funding Number: The Lundbeck Foundation)
Record Dates: First submitted 2020-04-13; First posted 2020-04-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid Plasma Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to examine the inflammatory response in the pulmonary compartment and blood of critically ill patients admitted to the ICU with COVID-19.

DETAILED DESCRIPTION:
The mechanisms of the ARDS-like respiratory failure observed in patients with COVID-19 are currently unknown, but may be related to a distinct local immune response within the lung. In the present study, we will examine the cellular and humoral pulmonary immune response in mechanically ventilated patients admitted to the ICU with COVID-19 by examining immune cell profiles, cytokine patterns, and the complement pathway in bronchoalveolar lavage fluid, and relate it to the concomitant systemic inflammatory response. We will examine the patients on day 1-3 and 7-9 after ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18y
* Mechanical ventilation
* Verified COVID-19 (throat swab or tracheal aspirate positive for SARS-CoV-2)
* ARDS according to the Berlin definition

Exclusion Criteria:

* Untreated malignant tachycardia or bradycardia
* Suspected or verified intracranial hypertension (ICP > 15 mmHg)
* Unilateral lung ventilation
* Severe non-correctable coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated COVID-19 patients with ARDS included within 3 days of ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
White blood cell counts | Day 0 (subsequent to study inclusion in the ICU)
  Total white blood cells, neutrocytes, lymphocytes, and monocytes in bronchoalveolar lavage fluid and blood
White blood cell counts | Day 7
  Total white blood cells, neutrocytes, lymphocytes, and monocytes in bronchoalveolar lavage fluid and blood
Lymphocyte populations | Day 0 (subsequent to study inclusion in the ICU)
  Cell populations and subpopulations evaluated by 10 colored flow cytometry (B cells, T cells, TCR subsets, Tregs/Th17, dendritic cells, myeloid cells and neutrophils) in bronchoalveolar lavage fluid and blood
Lymphocyte populations | Day 7
  Cell populations and subpopulations evaluated by 10 colored flow cytometry (B cells, T cells, TCR subsets, Tregs/Th17, dendritic cells, myeloid cells and neutrophils) in bronchoalveolar lavage fluid and blood

SECONDARY OUTCOMES:
Cytokines | Day 0 (subsequent to study inclusion in the ICU)
  Multiplex assay for measuring cytokines in bronchoalveolar lavage fluid and plasma (e.g. IL-1-beta, IL-1RA, IL-2, IL-6, IL-8, IL-10, IL-17, IL-18, IL-33, IL-35, TGF-beta, TNF-alpha, HMGB1)
Cytokines | Day 7
  Multiplex assay for measuring cytokines in bronchoalveolar lavage fluid and plasma (e.g. IL-1-beta, IL-1RA, IL-2, IL-6, IL-8, IL-10, IL-17, IL-18, IL-33, IL-35, TGF-beta, TNF-alpha, HMGB1)
Lectin complement pathway | Day 0 (subsequent to study inclusion in the ICU)
  MBL, ficolin-1, ficolin-2, ficolin-3, and MASPs in bronchoalveolar lavage fluid and plasma
Lectin complement pathway | Day 7
  MBL, ficolin-1, ficolin-2, ficolin-3, and MASPs in bronchoalveolar lavage fluid and plasma
Microorganisms | Up to 12 weeks
  Growth of pathogenic microorganisms in body fluids (e.g. urine, blood, bronchoalveolar lavage fluid)
Respiratory pathogens | Day 0 (subsequent to study inclusion in the ICU)
  Respiratory filmarray PCR for testing for pathogens
Respiratory pathogens | Day 7
  Respiratory filmarray PCR for testing for pathogens
Ribosomal RNA in the airways | Day 0 (subsequent to study inclusion in the ICU)
  16S ribosomal RNA (rRNA) and 18S rRNA PCR for bacterial or fungal pathogen identification in bronchoalveolar lavage fluid
Ribosomal RNA in the airways | Day 7
  16S ribosomal RNA (rRNA) and 18S rRNA PCR for bacterial or fungal pathogen identification in bronchoalveolar lavage fluid
Levels of SARS-CoV-2 in the airways | Day 0 (subsequent to study inclusion in the ICU)
  Semiquant PCR of SARS-CoV-2 in bronchoalveolar lavage fluid
Levels of SARS-CoV-2 in the airways | Day 7
  Semiquant PCR of SARS-CoV-2 in bronchoalveolar lavage fluid
Surfactant in the airways | Day 0
  Measured in bronchoalveolar lavage fluid by fourier-transform infrared spectroscopy using the dipalmitoylphosphatidylcholine[DPPC]/spingomyelin[SM]) ratio
Autoantibodies against type I IFNs in the airways | Day 0
  Measured in bronchoalveolarlavage fluid

OTHER OUTCOMES:
Mortality | Up to 6 months
  ICU mortality
Mortality II | Up to 6 months
  In hospital mortality
Blood markers of inflammation | Daily assessment in the ICU up to 12 weeks
  C-reactive protein, procalcitonin, ferritin
Infiltrates on conventional chest x-ray | Up to 12 weeks
  Number of participants with unilateral infiltrates or bilateral infiltrates and/or air bronchogram

CONTACTS AND LOCATIONS:
Overall Officials: Ronni R Plovsing, MD, PhD, Principal Investigator — Dept. of Intensive Care, University Hospital Hvidovre, Denmark
Locations (1):
- Dept. of Intensive Care 542, University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fahnoe U, Ronit A, Berg RMG, Jorgensen SE, Mogensen TH, Underwood AP, Scheel TKH, Bukh J, Plovsing RR. A Distinct Dexamethasone-Dependent Gene Expression Profile in the Lungs of COVID-19 Patients. J Infect Dis. 2022 Dec 13;226(12):2137-2141. doi: 10.1093/infdis/jiac218. PMID 35639922